CLINICAL TRIAL: NCT07058597
Title: Assessment of Mental Nerve Integrity During Fixation of Fractures at Anterior Transition Zone Using Three Different Miniplates Configurations
Brief Title: Fixation of Fractures at Anterior Transition Zone Using Three Different Miniplates Configurations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AMTZ-3G-2025
Record Dates: First submitted 2025-07-01; First posted 2025-07-10 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Mandibular Fracture Trauma; Mandible Fracture
Keywords: mandibular fractures; anterior transition zone; mental nerve; electrophysiological study
MeSH Terms: conditions — Mandibular Fractures

STUDY DESIGN:
Intervention Model Description: Patients with with fractures in the anterior transition zone managed with 3 different configurations of miniplates
Who Masked: Participant, Care Provider
Masking Description: Sequentially numbered, opaque, sealed envelopes (SNOSE) allocation concealment method will be utilized. Each participant included in the study will be given a serial number that will be used in the allocation. These numbers will be written in identical sheets of paper with the group to which each participant is allocated and placed inside opaque envelopes carrying the respective names of participants. A trial independent personnel will be assigned the role of keeping the envelopes and unfolding them only at the time of the operation, so that the participant is allocated to a group which is concealed from the operator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Patients with mandibular fracture in the anterior transition zone managed with Twinfork plate (Active Comparator): Patients with mandibular fracture in the anterior transition zone managed with Twinfork plate
  Interventions: Device: Twinfork plate
- Patients with mandibular fracture in the anterior transition zone managed with 3D-interlocking (Active Comparator): Patients with mandibular fracture in the anterior transition zone managed with 3D-interlocking plate
  Interventions: Device: 3D-interlocking plate
- Patients with mandibular fracture in the anterior transition zone managed with miniplates (Experimental): Patients with mandibular fracture in the anterior transition zone managed with miniplates
  Interventions: Device: Miniplate

INTERVENTIONS:
Device: Twinfork plate — Twinfork plate
  Arms: Patients with mandibular fracture in the anterior transition zone managed with Twinfork plate
Device: 3D-interlocking plate — 3D-interlocking plate
  Arms: Patients with mandibular fracture in the anterior transition zone managed with 3D-interlocking
Device: Miniplate — Miniplate
  Arms: Patients with mandibular fracture in the anterior transition zone managed with miniplates

SUMMARY:
Fractures involving the anterior transition zone of the mandible are frequently encountered and hold particular clinical significance due to the presence of the mental nerve. Consequently, mental nerve paresthesia is among the common postoperative complications associated with these fractures. To assess the mental nerve functional integrity during fixation of fractures at the anterior transition zone using twin fork-miniplate, 3d interlocking miniplate and two miniplates

DETAILED DESCRIPTION:
A total of 36 patients (they were divided into three groups 16 patients in each group ) with parasymphyseal-body fractures , one group was treated with twin-fork miniplate , the second group was treated using 3d interlocking miniplate and the third one was treated with conventional two miniplates. Postoperative evaluation of the mental nerve was conducted using both subjective and objective methods at intervals of 24 hours, and at 1, 4, 6 and 12 weeks. Furthermore, an electrophysiological study was performed at 6 weeks postoperatively to measure the mental nerve's amplitude, onset latency and conduction velocity

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from recent, uninfected and minimally displaced or unfavorable fractures at parasymphysis-body region of the mandible
* Adult patients from 20-40 years old with no gender predilection that agreed to present for follow-up visits for a minimum postoperative period of 3 months.
* A fracture that demands open reduction and internal fixation.
* The patient medically fit for general anesthesia.

Exclusion Criteria:

* Medically compromised patients contradicting operation.
* Pathological fracture.
* An old fracture.
* Completely edentulous patient.
* Patients with frank infection.
* Patients with a comminuted fracture.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
Sensory nerve function | 6 weeks
  Objective assessment by using a dental probe pressure to determine any sensory changes along the distribution of the mental nerve in comparison to the contralateral side (nociceptive method).

SECONDARY OUTCOMES:
Radiographic evaluation for fracture healing | 3 months
  Preoperative CT scan will be obtained, immediate CT scan will be used to assess the adequacy of fracture line reduction and fixation, and then another CT will be taken at 12th week to estimate the mean bone density at the fracture line in comparison with the immediate postoperative scan.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Alexandria University, Alexandria, Alexandria Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
all data will be de-identified to protect the participant data. patients signed an informed consent for the use of their medical records and data for study
Supporting Information: SAP
Access Criteria: to any one who required them after deidentification